CLINICAL TRIAL: NCT01713322
Title: Testing Educational Materials About Immunizations in a Paediatric Setting
Brief Title: Testing Educational Materials in a Paediatric Setting
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Anna Taddio, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-195C
Record Dates: First submitted 2012-10-21; First posted 2012-10-24 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Immunization
Keywords: parent education; pain management; immunization; infant
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pain management education (Experimental): Parents are provided with educational material on how to manage child pain during immunization.
  Interventions: Behavioral: Pain management education
- No pain management education (Other): Control - parents receive general information about childhood immunization.
  Interventions: Behavioral: No pain management education

INTERVENTIONS:
Behavioral: Pain management education — Parents are provided with educational material on how to manage child pain during immunization.
  Arms: Pain management education
Behavioral: No pain management education — Control - parents receive general information about childhood immunization.
  Arms: No pain management education

SUMMARY:
Immunization procedures are a common source of iatrogenic pain for infants. A recently developed clinical practice guideline, led by Taddio et al., created evidence-based strategies for management of immunization pain. User-friendly educational tools outlining these strategies were made. The goal of cluster randomized controlled trial is to assess whether these educational materials increase utilization of pain-relieving strategies by parents during infant immunizations.

DETAILED DESCRIPTION:
Immunization procedures are a common source of iatrogenic pain for infants. A recently developed clinical practice guideline led by Taddio et al. provides evidence-based recommendations for the management of immunization pain in children. User-friendly educational tools based on the guideline have also been developed, including a factsheet and educational video. The primary objective of this study is to assess whether these materials can increase utilization of pain -relieving strategies by parents during immunizations. Parents will be recruited during their infant's 2-month or 4-month scheduled visit to receive either the educational material related to immunization pain management (intervention group) or general information about immunization (control group). The study team will then follow these infants at their current and upcoming immunizations visit and document the pain management strategies utilized, infant pain responses, and parental satisfaction with pain management.

ELIGIBILITY:
Inclusion Criteria:

* Parents of 2 or 4-month old healthy infants during routine immunization appointments
* Parent accompanies infant at immunization appointments

Exclusion Criteria:

* Parents of infants <30 weeks gestational age (GA)
* Parents delaying infant immunization for >2 months
* Parents who are unable to read and understand English
* Infants with congenital anomalies, neurological conditions, and maternal psychiatric conditions

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Number of pain management strategies utilized | During immunization
  The number of pain management strategies utilized during immunization injections measured post-intervention from videotapes by a blinded assessor.

SECONDARY OUTCOMES:
Pain during infant immunizations | During immunization
  Pain during infant immunizations, as measured by a validated measure of pain in infants, the Modified Behavioural Pain Scale (MBPS), by trained and blinded research assistants.
Parent behaviour during infant immunizations | During immunization
  Parent behaviour during infant immunizations, as measured by Measure of Adult and Infant Soothing and Distress (MAISD) tool by trained and blinded research assistants.
Pain during infant immunizations as reported by parents | During immunization
  Pain during immunization appointments, as reported by parents using the Numerical Rating Scale (NRS), in real-time.
Parent-reported satisfaction with immunization experience | During immunization
  Parent-reported satisfaction with their immunization experience in their infant during immunization appointments on a 5-point Likert scale.
Duration of infant crying during immunizations | During immunization
  Duration of infant crying during infant immunizations, measured in seconds, will be assessed from videotapes by a trained and blinded assessor.
Pain during infant immunizations | During immunizations
  Pain during infant immunizations will be assessed by researchers, in real time, using the Numerical Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — University of Toronto
Locations (1):
- St. Michael's Health Center, Pediatric Clinic., Toronto, Ontario, Canada